CLINICAL TRIAL: NCT02930369
Title: A Randomized, Comparative, Prospective Study of Anatomical Outcomes With Different Internal Limiting Membrane Peeling Area in Surgery for Idiopathic Macular Hole
Brief Title: Effects of Different Area of Internal Limiting Membrane Peeling (ILM) Peeling on Anatomical Outcomes in Macular Hole Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Mingwei Zhao, Dr., Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAILMP-CHINA
Record Dates: First submitted 2016-10-10; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Macular Hole
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 4PD diameter of ILM peeling in surgery (Active Comparator): patients in this group was given 4papillary diameter (PD) diameter of internal limiting membrane (ILM) peeling in surgery
  Interventions: Procedure: ILM peeling surgery
- 2PD diameter of ILM peeling in surgery (Experimental): patients in this group was given 2PD diameter of ILM peeling in surgery
  Interventions: Procedure: ILM peeling surgery

INTERVENTIONS:
Procedure: ILM peeling surgery — 4PD or 2PD diameter of ILM peeling in surgery was given to patients with idiopathic macular hole (IMH)

SUMMARY:
The purpose of this study is to determine the effects of two different internal limiting membrane (ILM) peeling area on anatomical closure outcomes after macular hole surgery measured by optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

* patients with IMH
* patients signed the informed consent form (ICF)
* patients with course of IMH less than 3 years

Exclusion Criteria:

* patients with hyper myopia
* patients with traumatic macular hole
* accompanied or secondary of other fundus disease
* open or reopen after receiving MH surgery
* patients with retinal detachment
* received vitrectomy due to other diseases
* glaucoma cannot be controled by medication
* patients with other retinal or choroidal disease that may affect VA
* poor patients compliance
* poor condition that cannot undertake the surgery
* dioptric media opacities which make it difficult to exam fundus or measure on OCT

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-06; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Anatomical closure grades in OCT | 1 year

SECONDARY OUTCOMES:
Change of anatomical closure grades in OCT | 3 months, 6 months, 1 year
Change from baseline in BCVA (best corrected visual acuity) | 3 months, 6 months, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mingwei Zhao, M.D, Study Director — Peking University People's Hospital